CLINICAL TRIAL: NCT02605083
Title: A Phase 1-2 Dose Escalation and Cohort-Expansion Study of Oral eFT508 in Subjects With Advanced Solid Tumors
Brief Title: A Dose Escalation and Cohort-Expansion Study of Oral eFT508 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated after determination of the RP2D, prior to opening expansion cohorts)
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0001
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: Cancer; Neoplasm; Solid Tumor; Breast; Head and Neck; Lung; Pancreatic; Hepatic; Melanoma; Colon; Renal; Thyroid; Prostate; Ovarian; MNK1; MNK2; eIF4E
MeSH Terms: conditions — Neoplasms; Melanoma; Thyroid Diseases | interventions — tomivosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eFT508 (Experimental): Escalation cohort
  Interventions: Drug: eFT508

INTERVENTIONS:
Drug: eFT508 — Will be given orally once or twice daily. Each treatment cycle = 21 days.

SUMMARY:
This clinical trial is a Phase 1-2, open-label, sequential-group, dose-escalation and cohort-expansion study evaluating the safety, pharmacokinetics, pharmacodynamics, and antitumor activity of daily oral administration of eFT508.

DETAILED DESCRIPTION:
eFT508 is an oral, potent and highly selective inhibitor of mitogen-activated protein kinase interacting kinase (MNK) 1 and 2. Dysregulated translation of messenger RNA (mRNA) plays a role in the pathogenesis of multiple solid tumors and hematological malignancies. MNK1 and MNK2 integrate signals from several oncogenic and immune signaling pathways (including RAS, p38 and Toll-like receptors) by phosphorylating eukaryotic initiation of factor 4E (eIF4E) and key effector proteins. Phosphorylation of these regulatory proteins by MNK1 and MNK2 selectively regulates the stability and translation of a subset of cellular mRNA that control tumor growth, the tumor microenvironment and immune signaling. Nonclinical studies indicate that eFT508 shows activity against various types of solid tumors. These nonclinical studies support initiation of clinical development of eFT508 in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
2. Pathologically documented diagnosis of advanced solid tumor malignancy that progressed after appropriate prior therapy or has no potential for cure with currently available treatments.
3. Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) outside of any prior radiation field.
4. At least 3 weeks post any treatments/therapies at the time of first dose.
5. Adequate bone marrow function.
6. Adequate hepatic function.
7. Adequate renal function.
8. Normal coagulation panel.
9. Negative antiviral serology.
10. Willingness to use effective contraception.

Exclusion Criteria:

1. Known central nervous system malignancy.
2. Gastrointestinal disease that may interfere with drug absorption.
3. Significant cardiovascular disease.
4. Significant ECG abnormalities.
5. Ongoing risk of bleeding due to active peptic ulcer disease, bleeding diathesis, or requirement for systemic anticoagulants. Use of heparin or thrombolytic agents for local maintenance or clearance of a central venous catheter is permitted.
6. Ongoing systemic bacterial, fungal or viral infection (with the exception of fungal infections of the skin or nails).
7. Pregnancy or breastfeeding.
8. Major surgery within 4 weeks before the start of study therapy.
9. Prior solid organ or bone marrow progenitor cell transplantation.
10. Prior therapy with any known inhibitor of MNK1 or MNK2.
11. Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids (can be using topical or inhaled corticosteroids).
12. Use of drugs that might pose a risk of a drug-drug interaction within 4-7 days before the start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/Recommended dose (RD) | Up to one year
Overall response rate (ORR) | Up to three years

SECONDARY OUTCOMES:
Safety (Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE v. 4.03)) | Up to three year
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE v. 4.03)
Plasma concentration of eFT508 as characterized by maximum serum concentration (Cmax) | Different time points up to 336 hours
Plasma concentration of eFT508 as characterized by Area Under the Curve (AUC) | Different time points up to 336 hours
Changes in eIF4E phosphorylation in peripheral blood cells (PBMCs) | Up to Day 14
Tumor control evaluated by modified RECIST criteria v 1.1 | Up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — Effector Therapeutics
Locations (4):
- United States (4):
  - SCRI at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No